CLINICAL TRIAL: NCT02428114
Title: A Multi Centre Study to Determine the Feasibility of Using an Integrated Consent Model to Compare Standard of Care Administration Schedules of G-CSF (Filgrastim) for Primary Prophylaxis of Chemotherapy-Induced Febrile Neutropenia in Early Stage Breast Cancer (React-G Study)
Acronym: React-G
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: OTT 14-05
Record Dates: First submitted 2015-04-15; First posted 2015-04-28 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Early Stage Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 5 days of filgrastim: Standard of care
- 7 days of filgrastim: Standard of care
- 10 days of filgrastim: Standard of care

SUMMARY:
In patients with early-stage breast cancer, chemotherapy has substantially improved survival rates for breast cancer patients. Improvements in outcomes, however, are compromised by the considerable toxicities associated with chemotherapy, most notable being neutropenia. Neutropenia is the presence of abnormally few white blood cells, leading to increased susceptibility to infection and can require hospitalization and need for intravenous antibiotics and is sometimes fatal. Febrile neutropenia can also be associated with treatment delays and dose reductions, potentially compromising treatment efficacy. Patients can receive medication to reduce the risk of febrile neutropenia, such as Neupogen (Filgrastim) as a daily injection for 5, 7, or 10 days. Since there is genuine uncertainty amongst healthcare professionals as to which administration schedule of Neupogen is better, investigators are performing a randomized study in which patients are put into a group by chance to give participants one of three standards of Neupogen daily injection. Neupogen can cost approximately $200 per injection, so if a physician prescribes 10 days for 8 cycles of treatment this can cost $16,000 compared to a 5 day prescription which would cost half this. In addition to cost savings, many patients are not able to give themselves injections on a daily basis and require nursing resources which are utilized at high-cost. This study will use an "integrated consent model" that involves an "oral consent" rather than a written informed consenting process in order to increase the number of patients who may participate while performing a study at a lower cost. While determining the optimal treatment will improve patient comfort and acceptability, using the minimal safe duration of administration may also offer cost savings.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary breast cancer
* Planned to start docetaxel component of FEC-D or AC-D, or first cycle of; dose-dense AC-T, TC, FEC-D or TAC chemotherapy
* ≥19 years of age
* Able to provide verbal consent

Exclusion Criteria:

* Contraindication to Filgrastim

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed breast cancer patients, who will be receiving FEC-D, AC-D, dose dense AC-T, TC or TAC chemotherapy will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of performing this study will be measured with composite endpoints: physician engagement, time for local or provincial research ethics approval, accrual rates, and patient/physician compliance. | 1 year

SECONDARY OUTCOMES:
Rates of documented febrile neutropenia (laboratory confirmation) | 1 year
ANC results at the end of each cycle of chemotherapy. | 1 year
hospital admissions | 1 year
percentage of patients who require chemotherapy dose delays | 1 year
percentage of patients who require chemotherapy dose decrease | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario

REFERENCES:
- [Derived] Clemons M, Fergusson D, Simos D, Mates M, Robinson A, Califaretti N, Zibdawi L, Bahl M, Raphael J, Ibrahim MFK, Fernandes R, Pitre L, Aseyev O, Stober C, Vandermeer L, Saunders D, Hutton B, Mallick R, Pond GR, Awan A, Hilton J. A multicentre, randomised trial comparing schedules of G-CSF (filgrastim) administration for primary prophylaxis of chemotherapy-induced febrile neutropenia in early stage breast cancer. Ann Oncol. 2020 Jul;31(7):951-957. doi: 10.1016/j.annonc.2020.04.005. Epub 2020 Apr 20. PMID 32325257
- [Derived] Ibrahim MFK, Hilton J, Mazzarello S, Fergusson D, Hutton B, Robinson A, Califaretti N, Hsu T, Gertler S, Mates M, Stober C, Vandermeer L, Mallick R, Clemons M. A multi-center pragmatic, randomized, feasibility trial comparing standard of care schedules of filgrastim administration for primary febrile neutropenia prophylaxis in early-stage breast cancer. Breast Cancer Res Treat. 2018 Apr;168(2):371-379. doi: 10.1007/s10549-017-4604-y. Epub 2017 Dec 6. PMID 29214415